CLINICAL TRIAL: NCT04927104
Title: Prospective, Single-arm, Single-center Exploratory Study on Safety of PEEK Knee Prosthesis
Brief Title: Exploratory Study on Safety of PEEK Knee Prosthesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Suzhou SinoMed Biomaterials Co., Ltd (Industry)
Responsible Party: Principal Investigator, You Wang, Prospective, Single-arm, Single-center Exploratory Study on Safety of PEEK Knee Prosthesis, RenJi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSSZZK2020001
Record Dates: First submitted 2021-06-10; First posted 2021-06-15 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Rheumatoid Arthritis of Knee; Osteoarthritis of the Knee
Keywords: TKA; PEEK Knee Prosthesis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: In this study, 10 subjects will be underwent total knee arthroplasty with PEEK knee prosthesis and be followed up 3, 6, and 12 months after surgery. The safety of the knee prosthesis for total knee arthroplasty will be investigated based on X-ray, magnetic resonance imaging, thin-section CT, hematological indexes, knee function, complications and the occurrence of serious adverse events at the 12-month follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEEK Knee Prosthesis (Experimental): In this study, 10 subjects will be underwent total knee arthroplasty with PEEK knee prosthesis.
  Interventions: Device: PEEK Knee Prosthesis

INTERVENTIONS:
Device: PEEK Knee Prosthesis — After subjects drop out of the study for any reason, the researchers can perform revision surgery using the prosthetic joint that is now routinely used.

SUMMARY:
In this study, 10 subjects will be underwent total knee arthroplasty with PEEK knee prosthesis and be followed up 3, 6, and 12 months after surgery. The safety of the knee prosthesis for total knee arthroplasty will be investigated based on X-ray, magnetic resonance imaging, thin-section CT, hematological indexes, knee function, complications and the occurrence of serious adverse events at the 12-month follow-up.

DETAILED DESCRIPTION:
According to the involved person's biomedical research ethics review method "(national health and family planning commission (11)) and the medical and health institutions to carry out the researchers launched a clinical research management method" (draft) on request, for national key development plan required for research and development production of PEEK knee prosthesis for clinical trials. In this study, 10 subjects will be underwent total knee arthroplasty with PEEK knee prosthesis and be followed up 3, 6, and 12 months after surgery. The safety of the knee prosthesis for total knee arthroplasty will be investigated based on X-ray, magnetic resonance imaging, thin-section CT, hematological indexes, knee function, complications and the occurrence of serious adverse events at the 12-month follow-up.

Since this study is an exploratory study, all subjects will be retrospectively studied one year after the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 55 years of age or older and less than 74 years of age, younger subjects should have urgent need for surgery.
* Subjects skeletal maturity.
* Subjects appropriate for total knee replacement, such as noninflammatory degenerative joint diseases (such as osteoarthritis, traumatic arthritis, or ischemic necrosis); Inflammatory degenerative joint diseases (including rheumatoid arthritis); Correction of functional deformity.
* The diseased side knee appropriate for primary total knee arthroplasty .
* Subjects or guardian is willing and able to sign the informed consent form .

Exclusion Criteria:

* Subjects with knee instability or abnormal gait caused by neuromuscular insufficiency.
* Subjects with bilateral knee joint disease who are expected to require replacement of both knees during the course of the study (i.e., within the next 12 months) .
* Alcoholics, drug addicts and drug abusers.
* Subjects with severe diabetes (fasting blood glucose > 10mmol/L)
* Body Mass Index, BMI>35.
* Female subjects who are pregnant or lactating.
* Subjects have disease limited their participation in the investigation or have an existing condition that would compromise their participation and follow-up in this clinical investigation.
* In the month before inclusion, subjects who participated in clinical studies of other drugs, biological agents or medical devices and failed to meet the main research endpoints.
* Other conditions, in the opinion of the Investigator, are inappropriate for participation in this clinical investigation.

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety measures at 12 months after surgery | 12 months
  The expected incidence of device-related complications within 12 months after surgery is 0.

SECONDARY OUTCOMES:
X-ray examination | At 3 and 12 months postoperatively
  At 3 and 12 months postoperatively, the prosthesis observed for clear lines and signs of loosening.
CT | one week and 12 months after surgery
  The wear of the prosthesis measured one week and 12 months after surgery.
MRI | 3 and 12 months after surgery
  Inflammation and effusion around the prosthesis assessed 3 and 12 months after surgery.
Hematological examination indexes 3 and 12 months after surgery | 3 and 12 months after surgery
  Including: blood routine, liver and kidney function, erythrocyte sedimentation rate, C-reactive protein
Excellent and good rates of the KSS knee scoring system at 3,6, 12 months postoperatively | 3,6, 12 months after surgery
  The full score of KSS is 100, above 85 is excellent, 70-84 is good, 60-69 is acceptable, and less than 60 is poor. Calculate the proportion of excellent and good grades.

OTHER OUTCOMES:
Incidence of other complications | 3,6, 12 months after surgery
  These include infection, knee stiffness, venous thrombosis in the lower extremities, and pulmonary embolism.

CONTACTS AND LOCATIONS:
Overall Officials: You Wang, MD, Principal Investigator — RenJi Hospital; Teng Long, MD, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital，Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT04927104/ICF_000.pdf